CLINICAL TRIAL: NCT00847743
Title: Effects of Tart Cherry Juice on Oxidative Stress and Inflammation in Older Men and Women
Brief Title: Study on Whether Tart Cherry Juice Can Reduce Oxidative Stress and Inflammation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kronos Longevity Research Institute (Other)
Collaborators: Vanderbilt University (Other)
Responsible Party: Tinna Traustadóttir, Ph.D., Kronos Longevity Research Institute
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: KLRI-2007-03
Record Dates: First submitted 2009-02-17; First posted 2009-02-19 (Estimated); Last update posted 2009-02-19 (Estimated); Status verified 2009-02

CONDITIONS: Oxidative Stress; Antioxidant Capacity; Inflammation
Keywords: oxidative stress; aging; ischemia-reperfusion
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Dietary Supplement: Tart Cherry Juice — 8 fl.oz. twice per day
  Other Names: CherryPharm

SUMMARY:
Oxidative stress has been linked to many diseases associated with aging, including coronary heart disease and Alzheimer's disease. Antioxidants and special proteins in the body work together to help prevent damage by free radicals. Some studies have indicated that as people age, they are less able to fight off oxidative stress and have increased levels of inflammation.

Tart cherries are known to be rich in antioxidants and plant-nutrients. The product we are using in this study is an all-natural tart cherry juice, mixed with apple juice concentrate and containing no additives and no preservatives.

We hope to learn whether antioxidant supplementation, such as tart cherry juice, can measurably decrease oxidative damage and inflammation associated with aging.

DETAILED DESCRIPTION:
Objectives

The primary objective of this pilot study is to investigate whether tart cherry juice consumption can reduce oxidative stress in older adults as measured by attenuation of F2-isoprostane responses to a forearm ischemia-reperfusion, and a decrease in urinary excretion products of oxidative damage. The secondary objective is to examine whether age-sensitive markers of inflammation are reduced in response to the cherry juice consumption.

ELIGIBILITY:
Inclusion Criteria:

* men and women, ages 55-80y, in good health, with >8 years of education
* non-smoker
* able to give informed consent

Exclusion Criteria:

* use of anti-oxidant supplements, in excess of a standard multi-vitamins
* current hormone replacement therapy
* any history of significant chronic disease
* uncontrolled hypertension
* body mass index (BMI) > 30 kg/m2
* high physical activity level, as determined by questions on the screening questionnaire
* use of anti-inflammatory medication

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-10; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
plasma F2-isoprostane response to a forearm ischemia-reperfusion challenge.

SECONDARY OUTCOMES:
Urinary markers of oxidative damage.

CONTACTS AND LOCATIONS:
Overall Officials: Tinna Traustadottir, Ph.D., Principal Investigator — Kronos Longevity Research Institute
Locations (1):
- Kronos Longevity Research Institute, Phoenix, Arizona, United States

REFERENCES:
- [Derived] Traustadottir T, Davies SS, Stock AA, Su Y, Heward CB, Roberts LJ 2nd, Harman SM. Tart cherry juice decreases oxidative stress in healthy older men and women. J Nutr. 2009 Oct;139(10):1896-900. doi: 10.3945/jn.109.111716. Epub 2009 Aug 19. PMID 19692530